CLINICAL TRIAL: NCT01770639
Title: A Retrospective Study to Assess the Outcome After Surgical Reconstruction of the Midfoot With the Midfoot Fusion Bolt in Patients With Neuroarthropathy
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: MFB Retro
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Charcot Neuroarthropathy; Diabetic Foot
Keywords: charcot foot; charcot neuroarthropathy; midfoot arthrodesis; midfoot fusion
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MFB: Surgical arthrodesis of the midfoot with the Midfoot Fusion Bolt (MFB)
  Interventions: Procedure: MFB

INTERVENTIONS:
Procedure: MFB — Surgical arthrodesis of the midfoot with the Midfoot Fusion Bolt (MFB)

SUMMARY:
The aim of this study is to investigate the clinical outcomes of surgical correction of foot deformity with the MFB in a larger group of patients with neurological impairment of the foot.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 at date of inclusion
* Previous surgical reconstruction of the midfoot with Midfoot Fusion Bolt(s) for one of the following indications:

Neuroarthropathy Deformity of the foot with neurological impairment - Signed informed consent according to local regulation

Exclusion Criteria:

- Prisoner at date of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuro-osteoarthropathy of the foot or with other neurological impairment in combination with foot deformity who have previously undergone surgical reconstruction of the midfoot with the Midfoot Fusion Bolt.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Treatment failure within the first year after surgery | Date of surgery to 1 year posto-op
  The occurrence and the date of a secondary surgical intervention for correction of deformity or an amputation within the first year after surgery.

SECONDARY OUTCOMES:
Treatment failure within the first two years after surgery | Date of surgery to 2 years post-op
  The occurrence and the date of a secondary surgical intervention for correction of deformity or an amputation within the first two years after surgery.
Adverse events related to the treatment or device under investigation | Date of surgery to 2 years post-op
  The occurrence, type, and date of adverse events related to the midfoot arthrodesis or the MFB within the first two years after surgery.
Immobilization and non-weightbearing | Date of surgery to time of full weightbearing
  The duration and type of postoperative immobilization and the duration of postoperative non-weightbearing.
Surgery details | Date of surgery
  Technical details of the midfoot reconstruction surgery .
Foot angles | Pre-op, post-op, 6w, 12w, 6m, 12m
  Talus-first metatarsal angle and calcaneus-fifth metatarsal angle on the AP and lateral x-rays of the affected foot before surgery, immediately after surgery, 6 weeks, 12 weeks, 6 months, and 12 months after surgery.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Universitätsklinikum Dresden, Dresden
  - Universität Rostock, Rostock
  - Klinik für Fuss und Sprunggelenkchirurgie Rummelsberg, Rummelsberg

REFERENCES:
- [Derived] Richter M, Mittlmeier T, Rammelt S, Agren PH, Hahn S, Eschler A. Intramedullary fixation in severe Charcot osteo-neuroarthropathy with foot deformity results in adequate correction without loss of correction - Results from a multi-centre study. Foot Ankle Surg. 2015 Dec;21(4):269-76. doi: 10.1016/j.fas.2015.02.003. Epub 2015 Mar 9. PMID 26564730